CLINICAL TRIAL: NCT02957357
Title: Optimizing the Effectiveness of Routine Post-treatment Surveillance in Prostate Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AFT-30
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-05

CONDITIONS: Cancer of Prostate; Cancer of the Prostate; Prostate Cancer; Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- National Cancer Data Base: Patients within the National Cancer Database with newly diagnosed prostate cancer between 2004 and 2010. Participating institutions each provided a random of sample of 10 patients to be included in the final cohort.
- NC ProCESS: The North Carolina Prostate cancer Comparative Effectiveness & Survivorship Study (NC ProCESS) is a prospective population-based cohort of >1,000 patients with newly diagnosed prostate cancer, enrolled from January 2011 through June 2013.

SUMMARY:
Through this study, the investigators seek to identify the benefits (improved survival) and harms (more procedures, more treatment, side effects, and quality-of-life impact) from different surveillance frequencies-every three vs. six vs. 12 months. Using the National Cancer Database and quality-of-life data from a large group of prostate cancer survivors, the investigators aim to compare survival, procedures/tests, treatments, and side effects in prostate cancer survivors who are followed with alternative surveillance frequencies and compare quality-of-life outcomes. The overall goal of the study is to provide high-quality data that will allow development of a personalized, risk-based tailored approach to post-treatment surveillance for prostate cancer.

DETAILED DESCRIPTION:
We seek to identify the benefits (improved survival) and harms (more procedures, more treatment, side effects, and quality-of-life impact) from different surveillance frequencies--every three vs. six vs. 12 months. We hypothesize that patients with a low risk of recurrence may experience more harm than benefit, while patients with a high risk of recurrence may have improved survival from frequent surveillance.

Specific aims: The specific aims are 1) compare survival, procedures/tests, treatments, and side effects in prostate cancer survivors who are followed with alternative surveillance frequencies; and 2) compare quality-of-life outcomes.

Methods:

Aim 1 will use the National Cancer Database, which includes 70 percent of cancer patients across the United States, and will provide results representative of outcomes of prostate cancer survivors. We will compare the effectiveness of the three most common surveillance frequencies (PSA testing every 3 months vs. 6 months vs. 12 months) stratified by risk of recurrence (low-risk, intermediate-risk, high-risk; as defined by the National Comprehensive Cancer Network (NCCN)) and initial treatment (surgery or radiation). The objective of this aim is to quantify the potential benefits (survival) and harms (procedures/tests, treatments, morbidity consequences) of different PSA surveillance frequencies in the 6 patient groups.

The objective of Aim 2 is to quantify the impact of different surveillance frequencies from the patient's perspective. This aim will use quality-of-life data from the North Carolina Prostate cancer Comparative Effectiveness & Survivorship Study (NC ProCESS), PI Ronald Chen, a prospective population-based cohort of >1,000 patients with newly diagnosed prostate cancer, enrolled from January 2011 through June 2013. Comparison groups are the same as Aim 1. PSA frequency will be similarly defined using medical record abstraction.

Patient and stakeholder engagement: Through a five-year process, patients have worked with the PI in all phases of this research, including 1) identifying the highest priority research topic, 2) defining the study population/comparators, and 3) identifying outcomes of highest relevance to patients. Patients and other stakeholders will continue to 4) monitor study conduct and progress and 5) design dissemination activities.

ELIGIBILITY:
Inclusion Criteria for the National Cancer Data Base cohort:

* Patient data part of the NCDB
* Diagnosed with prostate cancer in 2004-2005.
* Treated for prostate cancer with surgery (prostatectomy) or radiation therapy

Inclusion/Exclusion Criteria for the NC ProCESS cohort:

Inclusion Criteria:

* Newly-diagnosed, histologically-proven, localized prostate adenocarcinoma.
* Completion of baseline interview prior to initiating therapy.
* Patient ability to complete study interview: no cognitive impairment, language or hearing problems.
* Not diagnosed with prostate cancer through transurethral resection of the prostate (TURP).
* Age 35-80.
* English speaking.
* Has telephone.

Exclusion Criteria:

* Initiation of treatment for prostate cancer prior to completion of baseline interview.
* Cognitive impairment.
* Hearing problems.
* Inability to speak or understand English.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 14,000 prostate cancer patients in the National Cancer Data Base (nationwide cancer registry) will be analyzed.
  The investigators will analyze data from the National Cancer Data Base (NCDB), a cancer registry which is maintained by the American College of Surgeons Commission on Cancer (CoC). Cancer registry staff review hospital and provider records to collect necessary data for the cancer registry so data are available for analysis for this project. There are >1400 CoC-hospitals; 10 patients will be sampled at each hospital thus 14,000 patients will be available for analysis.
  The NC ProCESS cohort consists of newly-diagnosed, early stage (localized, non-metastatic) prostate cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 11314 (Actual)
Dates: Start 2016-02; Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Chen, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share data or to make individual participant data available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | National Cancer Data Base | NC ProCESS
Started | 10479 | 835
Completed | 10479 | 835
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | National Cancer Data Base | NC ProCESS | Total
Number analyzed (Participants) | 10479 | 835 | 11314
Age, Customized [Count of Participants; unit: Participants]
  Age group: <55 | 1329 | 115 | 1444
  Age group: 55-64 | 4059 | 334 | 4393
  Age group: 65-75 | 5091 | 345 | 5436
  Age group: >75 | 0 | 41 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10479 | 835 | 11314
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 7561 | 550 | 8111
  Non-Hispanic Black | 1375 | 248 | 1623
  Other | 1543 | 37 | 1580
Region of Enrollment [Number; unit: participants]
  United States | 10479 | 835 | 11314

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time to death or date of last follow-up after primary treatment with surgery or radiation.
Time Frame: From completion of primary treatment with surgery or radiation to the earliest occurrence of death, loss to follow-up, or the end of the study period.
Population: Analysis population comprised patients in the National Cancer Data Base, stratified by risk group (low, intermediate, high) and treatment (radiation or surgery). Survival data on patients in NC ProCESS were not collected for this assessment.
Measure: Median (Full Range); unit: years
Groups:
- Low Risk/Radiation: Patients with low-risk prostate cancer treated with radiation therapy
- Low Risk/Surgery: Patients with low risk prostate cancer treated with radical prostatectomy (i.e. surgery)
- Intermediate Risk/Radiation: Patients with intermediate risk prostate cancer treated with radiation therapy
- Intermediate Risk/Surgery: Patients with intermediate risk prostate cancer treated with radical prostatectomy (i.e. surgery)
- High Risk/Radiation: Patients with high risk prostate cancer treated with radiation therapy
- High Risk/Surgery: Patients with high risk prostate cancer treated with radical prostatectomy (i.e. surgery)
Arm/Group | Low Risk/Radiation | Low Risk/Surgery | Intermediate Risk/Radiation | Intermediate Risk/Surgery | High Risk/Radiation | High Risk/Surgery
Number analyzed (Participants) | 1891 | 1772 | 1818 | 2311 | 1326 | 1336
years
  Participants with <= 1 PSA test in the first year after treatment: number analyzed (Participants) | 670 | 588 | 658 | 715 | 469 | 454
  Participants with <= 1 PSA test in the first year after treatment | 8.7 [2.4 to 12.5] | 8.8 [2.2 to 12.3] | 8.6 [1.2 to 12.5] | 9.0 [2.2 to 12.5] | 8.8 [2.4 to 12.4] | 8.9 [2.3 to 12.5]
  Participants with 2 PSA tests in the first year after treatment: number analyzed (Participants) | 669 | 447 | 604 | 575 | 409 | 302
  Participants with 2 PSA tests in the first year after treatment | 8.2 [2.5 to 12.6] | 8.4 [2.5 to 12.4] | 8.3 [2.3 to 12.74] | 8.7 [2.3 to 12.4] | 8.6 [0.5 to 12.3] | 8.6 [2.2 to 12.4]
  Participants with >=3 PSA tests in the first year after treatment: number analyzed (Participants) | 552 | 737 | 556 | 1021 | 448 | 580
  Participants with >=3 PSA tests in the first year after treatment | 8.2 [2.3 to 12.2] | 8.6 [2.1 to 12.3] | 8.3 [2.4 to 12.4] | 8.9 [2.2 to 12.2] | 8.36 [2.2 to 12.2] | 8.9 [2.4 to 12.6]

2. Primary Outcome: Prostate Cancer Anxiety
Description: Prostate cancer anxiety was measured annually (starting 12 months after participant enrollment) using the validated Memorial Anxiety Scale for Prostate Cancer (MAX-PC). The instrument contains 18 questions across 3 subscales assessing anxiety related to prostate cancer (11 items), PSA testing (3 items), and fear of recurrence (4 items). Each item was scored on a Likert-type scale (1 to 4), with a higher score indicating greater anxiety. The subscale means represent the average scores across the items in that sub-scale. The mean Total MAX-PC scores represent the average scores across the 3 subscales (anxiety related to prostate cancer; anxiety related to PSA testing; and anxiety related to prostate cancer recurrence).
Time Frame: 12 to 60 months after participant enrollment
Population: The analysis population comprised participants from the North Carolina Prostate Cancer Comparative Effectiveness & Survivorship Study who received primary treatment with either radiation therapy or surgery.
  Data were not collected from the National Cancer Data Base for this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- <= 1 PSA Test in Year 1 After Treatment: Participants in the North Carolina Prostate Cancer Comparative Effectiveness & Survivorship Study who received primary treatment with radiation therapy or surgery and <=1 PSA tests in the first year after treatment.
- 2 PSA Tests in Year 1 After Treatment: Participants in the North Carolina Prostate Cancer Comparative Effectiveness & Survivorship Study who received primary treatment with radiation therapy or surgery and 2 PSA tests in the first year after treatment.
- >= 3 PSA Tests in Year 1 After Treatment: Participants in the North Carolina Prostate Cancer Comparative Effectiveness & Survivorship Study who received primary treatment with radiation therapy or surgery and >=3 PSA tests in the first year after treatment.
Arm/Group | <= 1 PSA Test in Year 1 After Treatment | 2 PSA Tests in Year 1 After Treatment | >= 3 PSA Tests in Year 1 After Treatment
Number analyzed (Participants) | 97 | 183 | 309
score on a scale
  Prostate Cancer Anxiety (Subscale 1) at 12 months | 1.56 (0.70) | 1.60 (0.74) | 1.52 (0.62)
  Prostate Cancer Anxiety (Subscale 1) at 24 months: number analyzed (Participants) | 73 | 173 | 296
  Prostate Cancer Anxiety (Subscale 1) at 24 months | 1.35 (0.57) | 1.57 (0.70) | 1.45 (0.60)
  Prostate Cancer Anxiety (Subscale 1) at 48 months: number analyzed (Participants) | 61 | 141 | 258
  Prostate Cancer Anxiety (Subscale 1) at 48 months | 1.40 (0.44) | 1.51 (0.53) | 1.47 (0.55)
  Prostate Cancer Anxiety (Subscale 1) at 36 months: number analyzed (Participants) | 54 | 135 | 243
  Prostate Cancer Anxiety (Subscale 1) at 36 months | 1.40 (0.57) | 1.51 (0.64) | 1.46 (0.63)
  Prostate Cancer Anxiety (Subscale 1) at 60 months: number analyzed (Participants) | 52 | 130 | 225
  Prostate Cancer Anxiety (Subscale 1) at 60 months | 1.37 (0.64) | 1.47 (0.63) | 1.39 (0.61)
  PSA Test Anxiety (Subscale 2) at 12 months | 1.19 (0.55) | 1.22 (0.49) | 1.15 (0.39)
  PSA Test Anxiety (Subscale 2) at 24 months: number analyzed (Participants) | 73 | 173 | 296
  PSA Test Anxiety (Subscale 2) at 24 months | 1.10 (0.32) | 1.23 (0.53) | 1.13 (0.39)
  PSA Test Anxiety (Subscale 2) at 36 months: number analyzed (Participants) | 61 | 141 | 258
  PSA Test Anxiety (Subscale 2) at 36 months | 1.16 (0.39) | 1.25 (0.55) | 1.16 (0.41)
  PSA Test Anxiety (Subscale 2) at 48 months: number analyzed (Participants) | 54 | 135 | 243
  PSA Test Anxiety (Subscale 2) at 48 months | 1.10 (0.26) | 1.23 (0.51) | 1.16 (0.48)
  PSA Test Anxiety (Subscale 2) at 60 months: number analyzed (Participants) | 52 | 130 | 225
  PSA Test Anxiety (Subscale 2) at 60 months | 1.11 (0.30) | 1.19 (0.48) | 1.11 (0.34)
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 12 months | 1.70 (0.68) | 1.82 (0.69) | 1.71 (0.60)
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 24 months: number analyzed (Participants) | 73 | 173 | 296
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 24 months | 1.68 (0.63) | 1.78 (0.61) | 1.70 (0.66)
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 36 months: number analyzed (Participants) | 61 | 141 | 258
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 36 months | 1.60 (0.63) | 1.85 (0.73) | 1.68 (0.63)
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 48 months: number analyzed (Participants) | 54 | 135 | 243
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 48 months | 1.64 (0.58) | 1.73 (0.62) | 1.75 (0.71)
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 60 months: number analyzed (Participants) | 52 | 130 | 225
  Prostate Cancer Recurrence Anxiety (Subscale 3) at 60 months | 1.70 (0.70) | 1.77 (0.59) | 1.69 (0.65)
  Total MAX-PC (average of subscale means) at 12 months | 1.53 (0.59) | 1.59 (0.60) | 1.50 (0.49)
  Total MAX-PC (average of subscale means) at 24 months: number analyzed (Participants) | 73 | 173 | 296
  Total MAX-PC (average of subscale means) at 24 months | 1.38 (0.47) | 1.57 (0.55) | 1.45 (0.50)
  Total MAX-PC (average of subscale means) at 36 months: number analyzed (Participants) | 61 | 141 | 258
  Total MAX-PC (average of subscale means) at 36 months | 1.43 (0.51) | 1.57 (0.56) | 1.44 (0.49)
  Total MAX-PC (average of subscale means) at 48 months: number analyzed (Participants) | 54 | 135 | 243
  Total MAX-PC (average of subscale means) at 48 months | 1.40 (0.44) | 1.51 (0.53) | 1.47 (0.55)
  Total MAX-PC (average of subscale means) at 60 months: number analyzed (Participants) | 52 | 130 | 225
  Total MAX-PC (average of subscale means) at 60 months | 1.40 (0.53) | 1.49 (0.51) | 1.42 (0.49)

3. Secondary Outcome: Time to Prostate Cancer Recurrence
Description: Time to recurrence represents the period between completion of the first course of treatment (i.e., radiation or surgery) and the date of prostate cancer recurrence (if prostate cancer recurrence occurred).
Time Frame: Completion of primary treatment with surgery or radiation to earliest of prostate cancer recurrence, loss to follow-up, or end of study period
Population: Analysis population comprised patients in the National Cancer Data Base, stratified by risk group (low, intermediate, high) and treatment (radiation or surgery). Prostate cancer recurrence was assessed within each strata by PSA testing frequency. Recurrence data on patients in NC ProCESS were not collected for this assessment.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Low Risk/Radiation | Low Risk/Surgery | Intermediate Risk/Radiation | Intermediate Risk/Surgery | High Risk/Radiation | High Risk/Surgery
Number analyzed (Participants) | 1807 | 1713 | 1760 | 2238 | 1273 | 1292
years
  <= 1 PSA test: number analyzed (Participants) | 612 | 548 | 622 | 674 | 439 | 432
  <= 1 PSA test | 4.4 (2.9) | 3.2 (3.2) | 4.4 (2.8) | 3.3 (2.7) | 3.5 (2.7) | 2.7 (2.5)
  2 PSA tests: number analyzed (Participants) | 654 | 436 | 589 | 563 | 399 | 290
  2 PSA tests | 5.5 (2.4) | 2.8 (2.2) | 4.5 (2.4) | 3.2 (2.4) | 3.8 (2.2) | 3.2 (2.6)
  >= 3 PSA tests: number analyzed (Participants) | 541 | 729 | 549 | 1001 | 435 | 570
  >= 3 PSA tests | 4.8 (2.9) | 3.4 (2.6) | 3.9 (2.2) | 3.7 (2.4) | 4.1 (2.6) | 2.9 (2.3)

4. Secondary Outcome: Treatment for Prostate Cancer Recurrence
Description: Receipt of subsequent treatment when prostate cancer has recurred after primary treatment with either surgery or radiation.
Time Frame: as for outcome 3
Population: Analysis population comprised patients in the National Cancer Data Base with prostate cancer recurrence, stratified by risk group (low, intermediate, high) and treatment (radiation or surgery). Treatment for recurrence was assessed within each strata by PSA testing frequency. Data on patients in NC ProCESS were not collected for this assessment.
Measure: Number (95% Confidence Interval); unit: percentage of men with recurrence
Arm/Group | Low Risk/Radiation | Low Risk/Surgery | Intermediate Risk/Radiation | Intermediate Risk/Surgery | High Risk/Radiation | High Risk/Surgery
Number analyzed (Participants) | 98 | 108 | 210 | 380 | 268 | 447
percentage of men with recurrence
  <= 1 PSA test: number analyzed (Participants) | 38 | 32 | 62 | 103 | 81 | 139
  <= 1 PSA test | 63.2 [46.0 to 78.2] | 84.4 [67.2 to 94.7] | 74.2 [61.5 to 84.5] | 88.3 [80.5 to 93.8] | 72.8 [61.8 to 82.1] | 94.2 [89.0 to 97.5]
  2 PSA tests: number analyzed (Participants) | 28 | 23 | 67 | 95 | 99 | 94
  2 PSA tests | 71.4 [51.3 to 86.8] | 91.3 [72.0 to 98.9] | 77.6 [65.8 to 86.9] | 94.7 [88.1 to 98.3] | 83.8 [75.1 to 90.5] | 92.6 [85.3 to 97.0]
  >= 3 PSA tests: number analyzed (Participants) | 32 | 53 | 81 | 182 | 88 | 214
  >= 3 PSA tests | 68.8 [50.0 to 83.9] | 88.7 [77.0 to 95.7] | 72.8 [61.8 to 82.1] | 89.6 [84.2 to 93.6] | 83.0 [73.4 to 90.1] | 94.9 [91.0 to 97.4]

5. Secondary Outcome: Prostate Cancer-Specific Health-Related Quality of Life
Description: Prostate cancer-specific health-related quality of life was assessed using the validated and well-published Prostate Cancer Symptom Indices (PCSI). PCSI assesses treatment-related morbidity and includes scales that measure sexual, bowel, and urinary symptoms. Patient responses are converted to a score from 0 (no symptoms) to 100 (maximum symptoms). A higher score indicates greater morbidity and poorer organ system function. PCSI was assessed at baseline, 3 months, 12 months and annually thereafter.
Time Frame: 12 to 60 months after participant enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | <= 1 PSA Test in Year 1 After Treatment | 2 PSA Tests in Year 1 After Treatment | >= 3 PSA Tests in Year 1 After Treatment
Number analyzed (Participants) | 97 | 182 | 309
score on a scale
  Sexual dysfunction at 12-months: number analyzed (Participants) | 96 | 181 | 303
  Sexual dysfunction at 12-months | 70.7 (32.9) | 64.5 (34.5) | 68.9 (31.3)
  Sexual dysfunction at 24-months: number analyzed (Participants) | 72 | 168 | 295
  Sexual dysfunction at 24-months | 68.4 (31.5) | 63.8 (35.2) | 68.2 (32.6)
  Sexual dysfunction at 36-months: number analyzed (Participants) | 59 | 140 | 252
  Sexual dysfunction at 36-months | 69.4 (32.7) | 64.8 (32.9) | 67.5 (33.9)
  Sexual dysfunction at 48-months: number analyzed (Participants) | 52 | 133 | 239
  Sexual dysfunction at 48-months | 74.9 (29.6) | 64.2 (34.8) | 69.3 (33.7)
  Sexual dysfunction at 60-months: number analyzed (Participants) | 51 | 126 | 220
  Sexual dysfunction at 60-months | 75.4 (26.8) | 69.7 (32.8) | 66.0 (35.4)
  Urinary incontinence at 12-months: number analyzed (Participants) | 97 | 176 | 307
  Urinary incontinence at 12-months | 25.4 (26.6) | 22.3 (26.6) | 29.4 (27.1)
  Urinary incontinence at 24-months: number analyzed (Participants) | 72 | 171 | 294
  Urinary incontinence at 24-months | 22.9 (26.6) | 22.5 (24.1) | 29.1 (26.8)
  Urinary incontinence at 36-months: number analyzed (Participants) | 61 | 138 | 256
  Urinary incontinence at 36-months | 24.3 (25.6) | 23.5 (24.9) | 27.5 (27.1)
  Urinary incontinence at 48-months: number analyzed (Participants) | 53 | 135 | 240
  Urinary incontinence at 48-months | 21.1 (23.9) | 25.0 (25.2) | 29.5 (26.3)
  Urinary incontinence at 60-months: number analyzed (Participants) | 52 | 126 | 222
  Urinary incontinence at 60-months | 24.0 (23.1) | 26.6 (27.4) | 29.1 (26.3)
  Urinary obstruction/irritation at 12-months: number analyzed (Participants) | 96 | 181 | 306
  Urinary obstruction/irritation at 12-months | 24.9 (14.2) | 21.8 (14.0) | 21.8 (14.1)
  Urinary obstruction/irritation at 24-months: number analyzed (Participants) | 73 | 171 | 294
  Urinary obstruction/irritation at 24-months | 20.2 (11.3) | 20.4 (13.5) | 20.6 (13.7)
  Urinary obstruction/irritation at 36-months: number analyzed (Participants) | 61 | 138 | 257
  Urinary obstruction/irritation at 36-months | 21.4 (11.4) | 20.6 (12.8) | 19.9 (13.0)
  Urinary obstruction/irritation at 48-months: number analyzed (Participants) | 53 | 133 | 242
  Urinary obstruction/irritation at 48-months | 20.0 (11.1) | 20.4 (13.3) | 20.8 (13.2)
  Urinary obstruction/irritation at 60-months: number analyzed (Participants) | 52 | 128 | 226
  Urinary obstruction/irritation at 60-months | 21.3 (11.6) | 21.4 (14.2) | 19.5 (12.6)
  Bowel dysfunction at 12-months | 8.7 (12.4) | 7.6 (9.6) | 6.3 (9.0)
  Bowel dysfunction at 24-months: number analyzed (Participants) | 73 | 173 | 296
  Bowel dysfunction at 24-months | 7.6 (9.3) | 8.0 (12.4) | 5.7 (8.2)
  Bowel dysfunction at 36-months: number analyzed (Participants) | 61 | 140 | 258
  Bowel dysfunction at 36-months | 7.7 (9.9) | 6.8 (9.0) | 5.9 (9.4)
  Bowel dysfunction at 48-months: number analyzed (Participants) | 54 | 136 | 243
  Bowel dysfunction at 48-months | 6.8 (7.0) | 6.2 (8.6) | 5.5 (8.4)
  Bowel dysfunction at 60-months: number analyzed (Participants) | 52 | 130 | 225
  Bowel dysfunction at 60-months | 8.5 (10.9) | 6.8 (9.3) | 6.1 (9.0)

6. Secondary Outcome: Global Health-Related Quality of Life
Description: Global health-related quality of life was assessed using the validated Short-Form 12 (SF-12). The SF-12 survey consists of Likert response formats and assesses overall health, mental health, vitality, social functioning, and whether one's daily physical activities are limited by their health or pain. The SF-12 also includes four binary response (yes or no) questions that assess limitations in function due to physical and emotional health. The SF-12 provides a Mental Component Score and a Physical Component Score, each calculated using norm-based scoring, with a mean score of 50 and standard deviation of 10. A lower score indicates lower health-related quality of life. SF-12 was assessed at baseline, 3 months, 12 months and annually thereafter.
Time Frame: 12 to 60 months after participant enrollment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | <= 1 PSA Test in Year 1 After Treatment | 2 PSA Tests in Year 1 After Treatment | >= 3 PSA Tests in Year 1 After Treatment
Number analyzed (Participants) | 97 | 180 | 309
score on a scale
  Physical health score at 12-months | 48.0 (9.7) | 49.2 (9.1) | 49.9 (9.7)
  Physical health score at 24-months: number analyzed (Participants) | 73 | 171 | 296
  Physical health score at 24-months | 45.9 (10.5) | 48.2 (10.2) | 48.5 (9.8)
  Physical health score at 36-months: number analyzed (Participants) | 61 | 141 | 257
  Physical health score at 36-months | 48.2 (10.4) | 48.0 (10.7) | 48.7 (9.4)
  Physical health score at 48-months: number analyzed (Participants) | 54 | 135 | 242
  Physical health score at 48-months | 47.9 (9.1) | 47.6 (10.0) | 48.0 (10.5)
  Physical health score at 60-months: number analyzed (Participants) | 50 | 128 | 223
  Physical health score at 60-months | 45.8 (10.5) | 45.5 (10.9) | 47.5 (9.9)
  Mental health score at 12-months | 53.9 (8.0) | 54.1 (7.4) | 54.7 (8.1)
  Mental health score at 24-months: number analyzed (Participants) | 73 | 171 | 296
  Mental health score at 24-months | 53.2 (8.3) | 53.2 (9.4) | 55.1 (8.4)
  Mental health score at 36-months: number analyzed (Participants) | 61 | 141 | 257
  Mental health score at 36-months | 53.6 (9.5) | 53.8 (9.1) | 54.7 (8.5)
  Mental health score at 48-months: number analyzed (Participants) | 54 | 135 | 242
  Mental health score at 48-months | 52.4 (10.3) | 54.2 (8.5) | 55.2 (8.6)
  Mental health score at 60-months: number analyzed (Participants) | 50 | 128 | 223
  Mental health score at 60-months | 53.6 (9.5) | 54.7 (7.8) | 55.3 (8.1)

ADVERSE EVENTS:
Time Frame: Adverse Events not monitored/assessed
Description: All-Cause Mortality, serious, and other adverse events were not monitored/assessed.
Arm/Group | National Cancer Data Base | NC ProCESS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/57/NCT02957357/Prot_SAP_000.pdf